CLINICAL TRIAL: NCT02793674
Title: High-Flow Nasal Cannula Flow Titration and Effort of Breathing in the Pediatric Intensive Care Unit
Brief Title: HFNC Flow Titration and Effort of Breathing in the PICU
Acronym: HFNCandEOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Robinder Khemani, Principal Investigator, Children's Hospital Los Angeles
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-14-00239
Record Dates: First submitted 2016-06-03; First posted 2016-06-08 (Estimated); Results first posted 2018-08-02 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: High Flow Nasal Cannula
Keywords: effort of breathing; high flow nasal cannula; respiratory distress
MeSH Terms: conditions — Dyspnea

ARMS (2):
- Fisher & Paykel high flow nasal cannula (Other): All participants in the study were on one or two high flow nasal cannula (HFNC) delivery systems. All were measured on the Fisher & Paykel HFNC delivery system. The flow rate of the HFNC was adjusted to determine if there exists a change in their effort of breathing.
  Interventions: Device: Fisher & Paykel high flow nasal cannula
- Vapotherm high flow nasal cannula (Other): All participants in the study were on one or two high flow nasal cannula (HFNC) delivery systems. A subgroup was measured on the Vapotherm HFNC delivery system. The flow rate of the HFNC was adjusted to determine if there exists a change in their effort of breathing.
  Interventions: Device: Vapotherm high flow nasal cannula

INTERVENTIONS:
Device: Fisher & Paykel high flow nasal cannula — Measurements of effort of breathing will be obtained at flow rates of 0.5, 1.0, 1.5, and 2.0 L/kg/min. Adequate time will be allowed at each flow rate for stabilization of EOB and flow levels will be trialed in a random order, each being trialed for approximately 5 minutes.
  Arms: Fisher & Paykel high flow nasal cannula
Device: Vapotherm high flow nasal cannula — Measurements of effort of breathing will be obtained at flow rates of 0.5, 1.0, 1.5, and 2.0 L/kg/min. Adequate time will be allowed at each flow rate for stabilization of EOB and flow levels will be trialed in a random order, each being trialed for approximately 5 minutes.
  Arms: Vapotherm high flow nasal cannula

SUMMARY:
High-flow nasal cannula (HFNC) is a method of non-invasive respiratory support used to decrease the effort of breathing (EOB) in patients with a wide variety of respiratory diseases in the pediatric intensive care unit. While its use has shown association with decreased rates of mechanical ventilation, there is a paucity of data examining its direct effect upon objective measurements of EOB. This study will aim to evaluate objective measurements of EOB in response to different levels of HFNC support, characterize the natural course of respiratory diseases treated with HFNC, evaluate changes in EOB secondary to the administration of supplemental medical therapies used in conjunction with HFNC, and compare different physiologic metrics for quantifying EOB in patients on HFNC.

ELIGIBILITY:
Inclusion Criteria:

* All participants less than or equal to three years old admitted to the PICU placed on high flow nasal cannula will be considered eligible for the study.

Exclusion Criteria:

* Participants will be excluded if they have a corrected gestational age less than 37 weeks or contraindications to nasoesophageal catheter placement (nasopharyngeal or esophageal abnormalities) or RIP bands (abdominal wall defects such as omphalocele). Patients greater than three years of age will be excluded.

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Lee JH, Rehder KJ, Williford L, Cheifetz IM, Turner DA. Use of high flow nasal cannula in critically ill infants, children, and adults: a critical review of the literature. Intensive Care Med. 2013 Feb;39(2):247-57. doi: 10.1007/s00134-012-2743-5. Epub 2012 Nov 10. PMID 23143331
- [Background] McKiernan C, Chua LC, Visintainer PF, Allen H. High flow nasal cannulae therapy in infants with bronchiolitis. J Pediatr. 2010 Apr;156(4):634-8. doi: 10.1016/j.jpeds.2009.10.039. Epub 2009 Dec 29. PMID 20036376
- [Background] Schibler A, Pham TM, Dunster KR, Foster K, Barlow A, Gibbons K, Hough JL. Reduced intubation rates for infants after introduction of high-flow nasal prong oxygen delivery. Intensive Care Med. 2011 May;37(5):847-52. doi: 10.1007/s00134-011-2177-5. Epub 2011 Mar 3. PMID 21369809
- [Background] Wing R, James C, Maranda LS, Armsby CC. Use of high-flow nasal cannula support in the emergency department reduces the need for intubation in pediatric acute respiratory insufficiency. Pediatr Emerg Care. 2012 Nov;28(11):1117-23. doi: 10.1097/PEC.0b013e31827122a9. PMID 23114231
- [Background] Frizzola M, Miller TL, Rodriguez ME, Zhu Y, Rojas J, Hesek A, Stump A, Shaffer TH, Dysart K. High-flow nasal cannula: impact on oxygenation and ventilation in an acute lung injury model. Pediatr Pulmonol. 2011 Jan;46(1):67-74. doi: 10.1002/ppul.21326. Epub 2010 Nov 23. PMID 21171186
- [Background] Lavizzari A, Veneroni C, Colnaghi M, Ciuffini F, Zannin E, Fumagalli M, Mosca F, Dellaca RL. Respiratory mechanics during NCPAP and HHHFNC at equal distending pressures. Arch Dis Child Fetal Neonatal Ed. 2014 Jul;99(4):F315-20. doi: 10.1136/archdischild-2013-305855. Epub 2014 Apr 30. PMID 24786469
- [Background] Bellani G, Pesenti A. Assessing effort and work of breathing. Curr Opin Crit Care. 2014 Jun;20(3):352-8. doi: 10.1097/MCC.0000000000000089. PMID 24722059
- [Background] Bekhof J, Reimink R, Brand PL. Systematic review: insufficient validation of clinical scores for the assessment of acute dyspnoea in wheezing children. Paediatr Respir Rev. 2014 Mar;15(1):98-112. doi: 10.1016/j.prrv.2013.08.004. Epub 2013 Oct 11. PMID 24120749
- [Background] Klein M, Reynolds LG. Relief of sleep-related oropharyngeal airway obstruction by continuous insufflation of the pharynx. Lancet. 1986 Apr 26;1(8487):935-9. doi: 10.1016/s0140-6736(86)91043-3. PMID 2871240
- [Background] Collett PW, Perry C, Engel LA. Pressure-time product, flow, and oxygen cost of resistive breathing in humans. J Appl Physiol (1985). 1985 Apr;58(4):1263-72. doi: 10.1152/jappl.1985.58.4.1263. PMID 3988680
- [Background] KRIEGER I, WHITTEN CF. WORK OF RESPIRATION IN BRONCHIOLITIS. Am J Dis Child. 1964 Apr;107:386-92. doi: 10.1001/archpedi.1964.02080060388010. No abstract available. PMID 14109498
- [Background] Stokes GM, Milner AD, Groggins RC. Work of breathing, intra-thoracic pressure and clinical findings in a group of babies with bronchiolitis. Acta Paediatr Scand. 1981 Sep;70(5):689-94. doi: 10.1111/j.1651-2227.1981.tb05769.x. PMID 7324919
- [Background] Allen JL, Wolfson MR, McDowell K, Shaffer TH. Thoracoabdominal asynchrony in infants with airflow obstruction. Am Rev Respir Dis. 1990 Feb;141(2):337-42. doi: 10.1164/ajrccm/141.2.337. PMID 2137313
- [Background] Mayfield S, Bogossian F, O'Malley L, Schibler A. High-flow nasal cannula oxygen therapy for infants with bronchiolitis: pilot study. J Paediatr Child Health. 2014 May;50(5):373-8. doi: 10.1111/jpc.12509. Epub 2014 Feb 25. PMID 24612137
- [Background] Milesi C, Baleine J, Matecki S, Durand S, Combes C, Novais AR, Cambonie G. Is treatment with a high flow nasal cannula effective in acute viral bronchiolitis? A physiologic study. Intensive Care Med. 2013 Jun;39(6):1088-94. doi: 10.1007/s00134-013-2879-y. Epub 2013 Mar 14. PMID 23494016
- [Background] Rubin S, Ghuman A, Deakers T, Khemani R, Ross P, Newth CJ. Effort of breathing in children receiving high-flow nasal cannula. Pediatr Crit Care Med. 2014 Jan;15(1):1-6. doi: 10.1097/PCC.0000000000000011. PMID 24201859
- [Background] Ritchie JE, Williams AB, Gerard C, Hockey H. Evaluation of a humidified nasal high-flow oxygen system, using oxygraphy, capnography and measurement of upper airway pressures. Anaesth Intensive Care. 2011 Nov;39(6):1103-10. doi: 10.1177/0310057X1103900620. PMID 22165366
- [Background] Lampland AL, Plumm B, Meyers PA, Worwa CT, Mammel MC. Observational study of humidified high-flow nasal cannula compared with nasal continuous positive airway pressure. J Pediatr. 2009 Feb;154(2):177-82. doi: 10.1016/j.jpeds.2008.07.021. Epub 2008 Aug 30. PMID 18760803
- [Background] Glezen P, Denny FW. Epidemiology of acute lower respiratory disease in children. N Engl J Med. 1973 Mar 8;288(10):498-505. doi: 10.1056/NEJM197303082881005. No abstract available. PMID 4346164
- [Background] Hartling L, Bialy LM, Vandermeer B, Tjosvold L, Johnson DW, Plint AC, Klassen TP, Patel H, Fernandes RM. Epinephrine for bronchiolitis. Cochrane Database Syst Rev. 2011 Jun 15;(6):CD003123. doi: 10.1002/14651858.CD003123.pub3. PMID 21678340
- [Background] Gadomski AM, Scribani MB. Bronchodilators for bronchiolitis. Cochrane Database Syst Rev. 2014 Jun 17;2014(6):CD001266. doi: 10.1002/14651858.CD001266.pub4. PMID 24937099
- [Background] Numa AH, Williams GD, Dakin CJ. The effect of nebulized epinephrine on respiratory mechanics and gas exchange in bronchiolitis. Am J Respir Crit Care Med. 2001 Jul 1;164(1):86-91. doi: 10.1164/ajrccm.164.1.2008090. PMID 11435244
- [Background] Sanchez I, De Koster J, Powell RE, Wolstein R, Chernick V. Effect of racemic epinephrine and salbutamol on clinical score and pulmonary mechanics in infants with bronchiolitis. J Pediatr. 1993 Jan;122(1):145-51. doi: 10.1016/s0022-3476(05)83508-5. PMID 8419602
- [Background] Willson DF, Horn SD, Hendley JO, Smout R, Gassaway J. Effect of practice variation on resource utilization in infants hospitalized for viral lower respiratory illness. Pediatrics. 2001 Oct;108(4):851-5. doi: 10.1542/peds.108.4.851. PMID 11581435
- [Background] Green M, Brayer AF, Schenkman KA, Wald ER. Duration of hospitalization in previously well infants with respiratory syncytial virus infection. Pediatr Infect Dis J. 1989 Sep;8(9):601-5. doi: 10.1097/00006454-198909000-00007. PMID 2797955
- [Background] Wang EE, Law BJ, Stephens D. Pediatric Investigators Collaborative Network on Infections in Canada (PICNIC) prospective study of risk factors and outcomes in patients hospitalized with respiratory syncytial viral lower respiratory tract infection. J Pediatr. 1995 Feb;126(2):212-9. doi: 10.1016/s0022-3476(95)70547-3. PMID 7844667
- See also: Study Results: The Relationship between High Flow Nasal Cannula Flow Rate and Effort of Breathing in Children — http://dx.doi.org/10.1016/j.jpeds.2017.06.006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study screened patients admitted to the PICU during the study period (September 2014 to June 2016) who were <3 years of age and started on high flow nasal cannula by the clinical team.
Pre-assignment Details: Of the 54 patients who met eligibility criteria on screening, 39% (N=21) underwent high flow nasal cannula flow titrations and had effort of breathing measurements taken.
Groups:
- Fisher & Paykel (FP) HFNC: A subgroup of participants were placed exclusively on Fisher & Paykel (FP) high flow nasal cannula (HFNC) (N=9). The flow rate of the HFNC was adjusted to determine if there existed a change in their effort of breathing (EOB) at different conditions.
  Measurements of effort of breathing was obtained at flow rates of 0.5, 1.0, 1.5, and 2.0 L/kg/min. Adequate time was allowed at each flow rate for stabilization of EOB and flow levels were trialed in a random order, each for approximately 5 minutes.
- Vapotherm (VT) HFNC: A subgroup of patients (N=12) had flow titrations performed on both Fisher & Paykel (FP) and Vapotherm (VT) high flow nasal cannula (HFNC) delivery systems. The flow rate of the HFNC was adjusted to determine if there existed a change in their effort of breathing (EOB) at different conditions. These patients had flow titrations on both HFNC delivery systems performed to compare EOB on these two different HFNC delivery systems. With one exception, titrations were performed on FP first, then crossed over to VT.
  Measurements of effort of breathing was obtained at flow rates of 0.5, 1.0, 1.5, and 2.0 L/kg/min. Adequate time was allowed at each flow rate for stabilization of EOB and flow levels were trialed in a random order, each for approximately 5 minutes.
Period: Overall Study
Arm/Group | Fisher & Paykel (FP) HFNC | Vapotherm (VT) HFNC
Started | 9 | 12
Completed | 9 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fisher & Paykel (FP) HFNC: A subgroup was studied on Fisher & Paykel (FP) high flow nasal cannula (HFNC) exclusively (N=9). The flow rate of the HFNC was adjusted to determine if there existed a change in their effort of breathing (EOB) at different conditions.
  Measurements of effort of breathing was obtained at flow rates of 0.5, 1.0, 1.5, and 2.0 L/kg/min. Adequate time was allowed at each flow rate for stabilization of EOB and flow levels were trialed in a random order, each for approximately 5 minutes.
- Vapotherm (VT) HFNC: A subgroup was studied on Vapotherm (VT) high flow nasal cannula (HFNC) (N=12). These patients then crossed over to the other arm and had back-to-back titrations on both types of HFNC (FP and VT). The flow rate of the HFNC was adjusted to determine if there existed a change in their effort of breathing (EOB) at different conditions.
  Measurements of effort of breathing was obtained at flow rates of 0.5, 1.0, 1.5, and 2.0 L/kg/min. Adequate time was allowed at each flow rate for stabilization of EOB and flow levels were trialed in a random order, each for approximately 5 minutes.
- Total: Total of all reporting groups
Arm/Group | Fisher & Paykel (FP) HFNC | Vapotherm (VT) HFNC | Total
Number analyzed (Participants) | 9 | 12 | 21
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 15 [5 to 25] | 4 [2 to 6] | 6 [2 to 12]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 5 | 7 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity / Race: African-American | 0 | 2 | 2
  Ethnicity / Race: Hispanic | 6 | 9 | 15
  Ethnicity / Race: Not specified | 3 | 1 | 4
Weight [Median (Inter-Quartile Range); unit: kilograms] | 9 [6.4 to 11] | 6.5 [4.8 to 7] | 6.5 [5 to 9]
Respiratory Illness [Number; unit: participants]
  Bronchiolitis | 6 | 7 | 13
  Pneumonia | 2 | 0 | 2
  Other | 1 | 5 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Pressure-rate Product (PRP) as a Function of Increasing HFNC Flow Rate on Both Types of HFNC Delivery System (FP and VT)
Description: PRP is a validated objective metric of effort of breathing which is derived from the product of the peak-to-trough change in esophageal pressure (in cmH20) and the respiratory rate (breaths per minute).
  The percent change in PRP is derived from the quotient of the absolute PRP at increased HFNC flow rates (1.0, 1.5, and 2.0 L/kg/min) divided by the absolute PRP at a baseline HFNC flow rate (0.5 L/kg/min). Percent change in PRP was used because a) there was a large degree of heterogeneity in baseline absolute PRP values in our study population based upon patient size, disease severity, and time point of illness, and b) we allowed for repeated measures on the same patient which would bias absolute PRP values in favor of those who were measured more frequently.
  It was not pre-specified to compare the two different HFNC delivery systems.
Time Frame: median percent change in PRP over 5 minute measurement period
Population: For this outcome measure, the arms/groups were combined to include all patients enrolled in the study. This included the patients studied on FP only (n=9) and those studied on VT and FP both (n=12) for a total n=21.
Measure: Median (Inter-Quartile Range); unit: percent change in PRP
Groups:
- Percent Change in Pressure-Rate Product: All participants in the study were placed on high flow nasal cannula (HFNC). For this outcome, the median percent change in PRP was obtained for all titrations on both types of HFNC delivery system (FP and VT).
  The flow rate of the HFNC was adjusted to determine if there existed a change in their effort of breathing (EOB) at different conditions.
  Measurements of effort of breathing was obtained at flow rates of 0.5, 1.0, 1.5, and 2.0 L/kg/min. Adequate time was allowed at each flow rate for stabilization of EOB and flow levels were trialed in a random order, each for approximately 5 minutes.
Arm/Group | Percent Change in Pressure-Rate Product
Number analyzed (Participants) | 21
percent change in PRP
  Percent Change in PRP at 1.0 L/kg/min | -10 [-22 to 0]
  Percent Change in PRP at 1.5 L/kg/min | -20 [-35 to -3.5]
  Percent Change in PRP at 2.0 L/kg/min | -23 [-33 to -9.0]

2. Secondary Outcome: Pressure-rate Product (PRP) as a Function of Increasing HFNC Flow Rate on Both Types of HFNC Delivery System (FP and VT)
Description: PRP is a validated objective metric of effort of breathing which is derived from the product of the peak-to-trough change in esophageal pressure (in cmH20) and the respiratory rate (breaths per minute). These values were obtained from 5 minute flow titration periods. For this outcome, the PRP was obtained for all titrations on both types of HFNC delivery system (FP and VT).
  It was not pre-specified to compare the two different HFNC delivery systems.
Time Frame: median PRP over a 5 minute period
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: cmH20 * breaths/minute
Groups:
- Pressure-Rate Product: All participants in the study were placed on high flow nasal cannula (HFNC). or this outcome, the PRP was obtained for all titrations on both types of HFNC delivery system (FP and VT).The flow rate of the HFNC was adjusted to determine if there existed a change in their effort of breathing (EOB) at different conditions.
  Measurements of effort of breathing was obtained at flow rates of 0.5, 1.0, 1.5, and 2.0 L/kg/min. Adequate time was allowed at each flow rate for stabilization of EOB and flow levels were trialed in a random order, each for approximately 5 minutes.
Arm/Group | Pressure-Rate Product
Number analyzed (Participants) | 21
cmH20 * breaths/minute
  PRP at 0.5 L/kg/min | 824 [592 to 1252]
  PRP at 1.0 L/kg/min | 699 [461 to 1080]
  PRP at 1.5 L/kg/min | 596 [406 to 923]
  PRP at 2.0 L/kg/min | 594 [365 to 893]

3. Secondary Outcome: Phase Angle as a Function of Increasing HFNC Flow Rate on Both Types of HFNC Delivery System (FP and VT)
Description: Phase angle is a measure of asynchrony between thoracic and abdominal breathing compartments that has correlated with increased effort of breathing. It is derived by measuring the relative expansion of these two breathing compartments and describing the synchrony between them as an angle (theta). For this outcome, the phase angle was obtained for all titrations on both types of HFNC delivery system (FP and VT).
  It was not pre-specified to compare the two different HFNC delivery systems.
Time Frame: median phase angle over a 5 minute period
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: degrees
Groups:
- Phase Angle: The phase angle was measured at all flow titrations for all patients on both types of HFNC delivery systems (FP and VT). This is a measure of thoracoabdominal asynchrony and a proxy for effort of breathing.
Arm/Group | Phase Angle
Number analyzed (Participants) | 21
degrees
  0.5 L/kg/min | 61 [40 to 115]
  1.0 L/kg/min | 61 [38 to 120]
  1.5 L/kg/min | 68 [38 to 122]
  2.0 L/kg/min | 59 [34 to 138]

4. Secondary Outcome: Percent Change in Pressure-rate Product (PRP) From Baseline as a Function of Increasing HFNC Flow Rate, Comparing Different HFNC Delivery Systems
Description: For this outcome, a subgroup of patients (N=12) were examined who had PRP measurements obtained on two different HFNC delivery systems (Fisher & Paykel (FP) and Vapotherm (VT)) in back-to-back flow titration periods. With one exception, patients were first studied on the FP and then transitioned to the VT HFNC delivery system.
Time Frame: median PRP over a 5 minute period
Population: Percent change in PRP from baseline (of 0.5 L/kg/min) was measured at different flow rates (1.0, 1.5, and 2.0 L/kg/min) for patients who had flow titrations done on the two different HFNC delivery systems (Fisher & Paykel (FP) and Vapotherm (VT)).
Measure: Median (Inter-Quartile Range); unit: percent change in PRP
Groups:
- Fisher & Paykel HFNC Delivery System: This arm shows the outcome (the median of the percent change in PRP from baseline as a function of flow rate) for these patients when they were studied on the FP HFNC delivery system.
- Vapotherm HFNC Delivery System: This arm shows the outcome (the median of the percent change in PRP from baseline as a function of flow rate) for these patients when they were studied on the VT HFNC delivery system.
Arm/Group | Fisher & Paykel HFNC Delivery System | Vapotherm HFNC Delivery System
Number analyzed (Participants) | 12 | 12
percent change in PRP
  1.0 L/kg/min | -15 [-22 to -5] | -9 [-18 to 4]
  1.5 L/kg/min | -19 [-42 to -7] | -22 [-30 to 2]
  2.0 L/kg/min | -23 [-36 to -17] | -11 [-32 to 8]

5. Secondary Outcome: Percent Change in Pressure-rate Product (PRP) From Baseline as a Function of Increasing HFNC Flow Rate, Comparing Weight-Stratified Subgroups on Both Types of HFNC Delivery System (FP and VT)
Description: To assess the relationship between patient size and dose-response of HFNC flow rate, we compared subgroups stratified by weight (patients <8 kg and >8 kg). For this outcome, the median percent change in PRP was obtained for all titrations on both types of HFNC delivery system (FP and VT).
  It was not pre-specified to compare the two different HFNC delivery systems.
Time Frame: medain percent change in PRP over a 5 minute period
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent change in PRP from baseline
Groups:
- Less Than or Equal to 8 kg; Greater Than 8 kg: The percent change in Pressure-rate Product (PRP) from baseline as a function of increasing HFNC flow rate was analyzed comparing weight-stratified subgroups. This analysis looked at the first titration performed on the HFNC delivery system for patients less than or equal to 8 kg (12 patients, 20 episodes) and greater than 8 kg (9 patients, 12 episodes). This outcome was derived from flow titraitons on both types of HFNC delivery system (FP and VT).
Arm/Group | Less Than or Equal to 8 kg | Greater Than 8 kg
Number analyzed (Participants) | 12 | 9
percent change in PRP from baseline
  1.0 L/kg/min | -14 [-23 to 0] | -5 [-10 to 3]
  1.5 L/kg/min | -27 [-44 to -5] | -2 [-22 to 5]
  2.0 L/kg/min | -25 [-45 to -16] | -15 [-29 to -8]

6. Secondary Outcome: Maximum Percent Change in Pressure-rate Product (PRP) From Baseline as a Function of Increasing HFNC Flow Rate, Comparing Weight-Stratified Subgroups on Both Types of HFNC Delivery System (FP and VT)
Description: Exploratory analysis of patients by further stratified weight groupings (<5 kg, 5-8 kg, and >8 kg) was performed to determine the greatest observed benefit of HFNC flow titration in patients of different sizes. For this outcome, the maximum percent change in PRP was obtained for all titrations on both types of HFNC delivery system (FP and VT).
  It was not pre-specified to compare the two different HFNC delivery systems.
Time Frame: median of the maximum percent change in PRP over a 5 minute period
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percent
Groups:
- Maximum Percent Change in PRP From Baseline Stratified by Wt: This analysis looked at the largest decrease in PRP for all flow titrations for weight stratified subgroups. For this outcome, the maximum percent change in PRP was obtained for all titrations on both types of HFNC delivery system (FP and VT).
Arm/Group | Maximum Percent Change in PRP From Baseline Stratified by Wt
Number analyzed (Participants) | 21
percent
  <5 kg | -46 [-52 to -29]
  5-8 kg | -30 [-48 to -6]
  >8 kg | -17 [-33 to 6]

ADVERSE EVENTS:
Time Frame: 22 months
Groups:
- Fisher & Paykel (FP) High Flow Nasal Cannula: A subgroup was studied on Fisher & Paykel (FP) high flow nasal cannula (HFNC) exclusively (N=9). The flow rate of the HFNC was adjusted to determine if there existed a change in their effort of breathing (EOB) at different conditions.
- Vapotherm (VT) High Flow Nasal Cannula: A subgroup was studied on Vapotherm (VT) high flow nasal cannula (HFNC) (N=12). These patients then crossed over to the other arm and had back-to-back titrations on both types of HFNC (FP and VT). The flow rate of the HFNC was adjusted to determine if there existed a change in their effort of breathing (EOB) at different conditions.
Arm/Group | Fisher & Paykel (FP) High Flow Nasal Cannula | Vapotherm (VT) High Flow Nasal Cannula
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/12
Other Adverse Events (participants affected / at risk) | 0/21 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fisher & Paykel (FP) High Flow Nasal Cannula (N=21) | Vapotherm (VT) High Flow Nasal Cannula (N=12)
any adverse event (Product Issues) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes